CLINICAL TRIAL: NCT04993898
Title: Effects of Plyometric Training on Endurance and Explosive Strength in Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/00848 Haris Hassan
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — Plyometric Exercise; Warm-Up Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training with warm up and cool down (Experimental): Plyometric training will include following exercises.
  * Squat to Squat Jump
  * Lunge to Plyo Lunge
  * Step Jack to Star Jumps
  * Plank to Plyo Spider Lunge
  * Plank to Frogger
  Interventions: Other: Plyometric training with warm up and cool down
- Conventional training with warm up & cool down (Active Comparator): Conventional training will include following exercises.
  * Squats
  * Single leg squat
  * Cork hip lift
  * Press ups
  Interventions: Other: Conventional training with warm up & cool down

INTERVENTIONS:
Other: Plyometric training with warm up and cool down — These Include Squat to Squat Jump, Lunge to Plyo Lunge, Step Jack to Star Jumps, Plank to Plyo Spider Lunge, Plank to Frogger Frequency = 2 days per week for 2 weeks and then 4 days per week after 2nd week to 4th week Intensity =500 jumps Time = 30 min
  Other Names: These Squat to Squat Jump, Lunge to Plyo Lunge, Step Jack to Star Jumps, Plank to Plyo Spider Lunge, Plank to Frogger
  Arms: Plyometric training with warm up and cool down
Other: Conventional training with warm up & cool down — These include Squats, Single leg squat, Cork hip lift, Press ups, Normal warm-up time 15 min before game.
  Arms: Conventional training with warm up & cool down

SUMMARY:
This study will help to understand the effects of plyometric training on endurance and explosive strength in cricket players.

DETAILED DESCRIPTION:
It will consist of combination of plyometric training with warm up and cool down including Squat to Squat Jump, Lunge to Plyo Lunge, Step Jack to Star Jumps, Plank to Plyo Spider Lunge, Plank to Frogger Frequency = 2 days per week for 2 weeks and then 4 days per week after 2nd week to 4th week, Intensity =500 jumps, Time = 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Active Male cricket players, age between 18-30 years.
* Playing from last 6 months.
* Normal BMI athletes

Exclusion Criteria:

* History of trauma/injury in last 2 months.
* Playing for less than 6 months.
* Over-weighted or underweighted athletes
* Any co-morbidity
* Cardiorespiratory issues like asthma
* Hypertension or Diabetes
* Meniscus or ACL/PCL/LCL/MCL injured patient
* Ankle sprain in last 6 month

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Jump Height | 6-8 Weeks
  Vertical jump tests is used to measure lower limb explosive power by measuring the height a client is able to jump in centimetre (cm).
  Attempt to touch the wall at the highest point of the jump. The difference in distance between the standing reach height and the jump height is the score. The best of three attempts is recorded.
Endurance | 6-8 Weeks
  This test is used to measures endurance
Ballistic push up test | 6-8 Weeks
  This test is used to measure explosive strength for upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Karim, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Cricket clubs located in Islamabad and Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SAPARİA A, Firmansyah D, HANIF AS. Plyometric Training Methods and Hand Eye Coordination on Volleyball Smash Skills in Sport Education Students, Tadulako University. International e-Journal of Educational Studies. 4:167-75.
- [Background] Warpeha JM. Upper body plyometrics. NSCA's Performance Training Journal. 2005; 6:6-8.
- [Background] Saez de Villarreal E, Requena B, Izquierdo M, Gonzalez-Badillo JJ. Enhancing sprint and strength performance: combined versus maximal power, traditional heavy-resistance and plyometric training. J Sci Med Sport. 2013 Mar;16(2):146-50. doi: 10.1016/j.jsams.2012.05.007. Epub 2012 Jun 21. PMID 22727979
- [Background] Zemkova E, Hamar D. Sport-Specific Assessment of the Effectiveness of Neuromuscular Training in Young Athletes. Front Physiol. 2018 Apr 11;9:264. doi: 10.3389/fphys.2018.00264. eCollection 2018. PMID 29695970
- [Background] Phillips E, Davids K, Renshaw I, Portus M. Acquisition of expertise in cricket fast bowling: perceptions of expert players and coaches. J Sci Med Sport. 2014 Jan;17(1):85-90. doi: 10.1016/j.jsams.2013.03.005. Epub 2013 Apr 22. PMID 23619161
- [Background] Houghton LA, Dawson BT, Rubenson J. Effects of plyometric training on achilles tendon properties and shuttle running during a simulated cricket batting innings. J Strength Cond Res. 2013 Apr;27(4):1036-46. doi: 10.1519/JSC.0b013e3182651e7a. PMID 22739327
- [Background] Malisoux L, Francaux M, Nielens H, Theisen D. Stretch-shortening cycle exercises: an effective training paradigm to enhance power output of human single muscle fibers. J Appl Physiol (1985). 2006 Mar;100(3):771-9. doi: 10.1152/japplphysiol.01027.2005. Epub 2005 Dec 1. PMID 16322375
- [Background] Suresh MM, Sundar K. EFFECT OF RESISTANCE TRAINING ON SELECTED BIO MOTOR VARIABLES AMONG ENGINEERING COLLEGE MEN CRICKET PLAYERS.
- [Background] Cowan C. The prevalence of injuries in women's cricket and its relationship to training practices and physical conditioning: Stellenbosch: Stellenbosch University; 2006.
- [Background] Feros SA, Young WB, O'Brien BJ. Relationship Between Selected Physical Qualities, Bowling Kinematics, and Pace Bowling Skill in Club-Standard Cricketers. J Strength Cond Res. 2019 Oct;33(10):2812-2825. doi: 10.1519/JSC.0000000000002587. PMID 29702520
- [Background] Beato M, Bianchi M, Coratella G, Merlini M, Drust B. Effects of Plyometric and Directional Training on Speed and Jump Performance in Elite Youth Soccer Players. J Strength Cond Res. 2018 Feb;32(2):289-296. doi: 10.1519/JSC.0000000000002371. PMID 29176387